CLINICAL TRIAL: NCT03029351
Title: GLP-1 Receptor Agonist Therapy and Albuminuria in Patients With Type 2 Diabetes
Acronym: 1981
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: termination by sponsor
Sponsor: University at Buffalo (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Paresh Dandona, SUNY Distinguished Professor, University at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1981 GLP
Record Dates: First submitted 2017-01-20; First posted 2017-01-24 (Estimated); Results first posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-03

CONDITIONS: Type2 Diabetes; Kidney Diseases
Keywords: albuminuria; GLP-1 Receptor Agonist; Type 2 Diabetes
MeSH Terms: conditions — Kidney Diseases; Albuminuria; Diabetes Mellitus, Type 2 | interventions — Exenatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Exenatide extended release (Experimental): Exenatide extended release treatment for 1 year on albuminuria levels in T2DM patients with micro- and macroalbuminuria compared to placebo.
  Interventions: Drug: Exenatide Extended Release for Inj Susp 2 MG
- Placebo (Placebo Comparator): Placebo treatment for 1 year on albuminuria levels in T2DM patients with micro- and macroalbuminuria compared to Exenatide extended release.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Exenatide Extended Release for Inj Susp 2 MG — Exenatide extended release treatment weekly for 1 year in T2DM patients with micro- and macroalbuminuria
  Other Names: Bydureon
  Arms: Exenatide extended release
Drug: Placebo — placebo treatment weekly for 1 year in type 2 diabetes with micro-and macroalbuminuria
  Arms: Placebo

SUMMARY:
This is a prospective study to evaluate effect of Exenatide extended release treatment for 1 year on albuminuria levels in T2DM patients with micro- and macroalbuminuria compared to placebo.

DETAILED DESCRIPTION:
This is a prospective study to evaluate effect of Exenatide extended release treatment for 1 year on albuminuria levels in T2DM patients with micro- and macroalbuminuria compared to placebo. The similarities in baseline values between the study groups will be compared using appropriate parametric tests. Transformations of the data on order to meet statistical assumptions may be considered. All statistical analysis will be carried out using SPSS software (SPSS Inc, Chicago, Illinois) based on intention to treat principle. Data will be presented as mean±standard error. The primary endpoint of the study is the change from baseline in albuminuria level at weeks 12, 26, 39 and 56 following Exenatide extended release and placebo treatments. Fasting samples collected at weeks 0, 12, 26, 39 and 56 will be used for this assessment with values at week 0 considered as baseline. Changes from baselines form both drugs arms will be compared to those from the placebo arms in both the micro and macroalbuminuria groups. The statistical analysis will be done using mixed model for repeated measurement (MMRM) analysis with assigned α value of 0.05. Our preliminary data on retrospective analysis of the difference in albuminuria following GLP-1RA treatment for 2.5 yrs in T2DM patients with micro and macroalbuminuria show regression of albuminuria (UACR) by approximately 55mg/mg and 500mg/g (about 50% reduction), respectively. Conservatively estimating a difference in the change from baseline in albuminuria after 1 year between the Exenatide extended release and placebo groups (across both albuminuria groups) of 60mg/g, with standard deviation of no more than 91mg/g, a sample size of 38 patients per group should provide adequate power (beta = 0.2) to detect a significant difference (alpha = 0.05). Assuming a drop-out rate of 15% and 2:1 drug:placebo randomization ratio, 60 active and 30 control will be recruited for a total of 90 patients (rounded up). Patients will be enrolled based on a predetermined stratification according to the two albuminuria categories (micro and macro at 1:1 ratio) with 45 patients in each.

The secondary end points include the comparison of the changes in albuminuria based on baseline albuminuria category (micro or macro), creatinine clearance, Cystatin C, TGFβ, type I and IV collagen, CTGF, and fibronectin levels, the expression of SMAD3, SMAD4, NQO-1, GST-1P and HO-1, Nrf-2/keap-1 system activation between the Exenatide extended release and placebo groups and across albuminuria categories

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes for at least 1 year.
* Microalbuminuria for at least 6 months (UACR: 30-300 mg/g)
* Macroalbuminuria for at least 6 months (UACR: >300 mg/g)
* HbA1c of ≤10%
* Ages 18-65 years (inclusive of ages 18 and 65)
* On ARBs/ACEi for at >3months

Exclusion Criteria:

* Use of GLP-1 Receptor agonists or SGLT-2 inhibitors therapy in the last 3 months
* History or risk for pancreatitis (e.g., history of gallstones, alcohol abuse, and hypertriglyceridemia)
* Coronary event or procedure (myocardial infarction, unstable angina, coronary artery bypass, surgery or coronary angioplasty) in the previous 3 months
* Hepatic disease: Severe hepatic insufficiency and/or significant abnormal liver function defined as:

  1. Aspartate aminotransferase (AST) >3x upper limit of normal (ULN) and/or alanine aminotransferase (ALT) >3x ULN
  2. Total bilirubin >2.0 mg/dL (34.2 µmol/L)
  3. Positive serologic evidence of current infectious liver disease including Hepatitis B viral antibody IGM, Hepatitis B surface antigen and Hepatitis C virus antibody
  4. Liver function tests more than 3 times the upper limit of normal
* Renal impairment (serum eGFR <30 ml/min)
* HIV
* Inability to give informed consent
* History of gastroparesis
* History of medullary thyroid carcinoma or MEN 2 syndrome
* Alcoholism
* Hypertriglyceridemia (>500 mg/dl).
* Any other life-threatening, non-cardiac disease
* Uncontrolled hypertension (BP > 160/100 mm of Hg)
* Congestive Heart Failure class III or IV
* Use of an investigational agent or therapeutic regimen within 30 days of study
* Participation in any other concurrent clinical trial
* Pregnant or breastfeeding patients or females of childbearing age not on 2 forms of acceptable contraceptives.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-01-10 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Diabetes Endocrinology Research Center of WNY, Williamsville, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Exenatide Extended Release | Placebo
Started | 7 | 8
Completed | 4 | 5
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exenatide Extended Release | Placebo | Total
Number analyzed (Participants) | 7 | 8 | 15
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 62 (8) | 65 (9) | 64 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 4 | 5 | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Urinary Albuminuria Levels
Description: change from baseline in 24-hr urinary albuminuria (albumin/creatine) level at week 52 following Exenatide extended release OR placebo treatments
Time Frame: baseline and 52 weeks
Measure: Mean (Standard Error); unit: microgram/mg creatinine
Arm/Group | Exenatide Extended Release | Placebo
Number analyzed (Participants) | 5 | 5
microgram/mg creatinine | -32 (122) | -12 (132)

ADVERSE EVENTS:
Time Frame: 52 weeks
Arm/Group | Exenatide Extended Release | Placebo
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/8
Other Adverse Events (participants affected / at risk) | 0/7 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-12): https://cdn.clinicaltrials.gov/large-docs/51/NCT03029351/Prot_SAP_002.pdf